CLINICAL TRIAL: NCT07306312
Title: Psychological Predictors of Pain and Disability in Patients With Chronic Low Back Pain After Manual Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Prentzas, Principal Investigator, PhD candidate, Physiotherapy Department University of Thessaly, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10130/25/TFSKTH - 04/04/25
Record Dates: First submitted 2025-11-16; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Disability Physical; Manual Theapy
Keywords: pain; disability; manual therapy; low back pain; Pain Neuroscience Education; psychological factors; kinesiophobia; catastrophizing; anxiety; depression; self-efficacy
MeSH Terms: conditions — Low Back Pain; Pain; Kinesiophobia; Anxiety Disorders; Depression | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Experimental): Participants with low back pain will be treated with manual therapy based on Maitland's principles
  Interventions: Other: Manual therapy
- Manual therapy plus Pain Neuroscience Education (Active Comparator): Participants with low back pain will be treated with manual therapy based on Maitland's principles but before that, volunteers will be participated, in a Pain Neuroscience Education (PNE) program
  Interventions: Other: Manual therapy plus Pain Neuroscience Education

INTERVENTIONS:
Other: Manual therapy — Manual therapy based on Maitland's approach
  Arms: Manual therapy
Other: Manual therapy plus Pain Neuroscience Education — Manual therapy based on Maitland's approach with Pain Neuroscience Education
  Arms: Manual therapy plus Pain Neuroscience Education

SUMMARY:
Low back pain has been reported to cause more disability than any other musculoskeletal health condition worldwide. About eight out of ten people will experience back pain at least once in their lifetime. The parameters that are usually evaluated in a low back pain condition are pain, functional disability and range of motion of the lumbar spine. There are studies that associate psychological conditions (self-efficacy, kinesiophobia, catastrophology, depression, anxiety) with pain and functional disability in patients with low back pain. However, the ability of psychological factors to predict progression after a program of physical therapy or therapeutic methods is not well studied.

The main purpose of this study is to investigate the predictive potential of psychological factors in the improvement of pain and functional disability after a manual therapy physiotherapy program in patients with chronic low back pain. A secondary purpose is to investigate the predictive potential of psychological factors in the improvement of pain and functional disability following a program of Pain Neuroscience Education (PNE) in patients with chronic low back pain. In addition, as a secondary purpose, it will be to investigate the effect of combining manual therapy therapy with PNE compared to manual therapy alone in patients with chronic low back pain.

This study will involve 60 people aged 18-65 with chronic low back pain, who will be randomly divided by lots into 2 groups of 30 people. The 1st group (30 people) will be treated with manual therapy based on Maitland's principles (interview, evaluation, mobilization), without any use of physiotherapy machines, but with the use of personalized exercises. The 2nd group (30 people) will do the same as group 1 and additional volunteers will participate in before, in a training program in Pain Neuroscience Education (PNE). The total number of sessions that each volunteer will receive will be 6, the duration of each session will be about 45 minutes, the frequency of the sessions will be 2 times a week and the total duration of the intervention will be 3 weeks. The associations between psychological states and clinical characteristics (pain, disability and range of motion) will be carried out with the Pearson or Spearman correlation coefficient depending on whether the data are parametric or not. Multiple regression models will also be created with predictive factors for psychological states and a predictive variable for each of the clinical parameters. The significance level will be set to p=0.05.

DETAILED DESCRIPTION:
Sample A total of 60 people with chronic low back pain will participate in the study and will be divided by lot into two groups of 30 people. The statistical calculation of the sample was made in the following way. We have 5 predictive factors (self-efficacy, depression, kinesiophobia, catastrophism and anxiety) and one predictive factor. According to the regression model we will need 10 people for each variable (i.e. 50 people). However, since we will divide the individuals into 2 groups, in order to have statistical strength in the measurements that will be made, we will take 30 people in each group Participants will be taken through convenience sampling. Participation in the survey will be voluntary and all those who take part will sign a consent form, after detailed information through the information form.

Equipment and Materials The equipment that will be used to conduct the study includes: a) a special electric manual therapy bed, adjustable in height, with recline and hole for the face b) two inclinometers to measure the range of motion of the lumbar spine, c) a mechanical algometer for measuring the pain threshold of the lumbar spine, d) specific questionnaires.

Interventions In both intervention groups, manual therapy based on Maitland's principles (interview, evaluation, mobilization) will be applied without the use of physiotherapy machines, but with the use of therapeutic exercise. The physiotherapist who will apply the techniques is a certified therapist of manual therapy Maitland Concept with 8 years of experience in the application of the method. The number of sessions that each volunteer will receive will be 6, the duration of each session will be about 45 minutes, the frequency of sessions will be 2 times a week and the total duration of the intervention will be 3 weeks.

The International Federation of Orthopaedic Manipulative Physical Therapists (IFOMPT) defines orthopaedic manual physical therapy as: "a specialized area of physiotherapy for the management of neuromusculoskeletal disorders, based on clinical reasoning, using very specific therapeutic approaches, including manual techniques and therapeutic exercises. Orthopedic hand-held physiotherapy also includes, and is guided by, the available scientific and clinical data and the biopsychosocial context of each individual patient".

The effectiveness of manual therapy in the treatment of low back pain (LBP) has been supported by various studies, indicating its potential benefits in reducing pain, improving impotence and trajectory range. Manual therapy includes techniques such as manipulation and mobilization, which have shown positive results in enhancing range of motion and relieving discomfort in patients with low back pain.

Treating low back pain through exercise has been shown to be an effective intervention, with various studies highlighting its benefits in reducing pain and improving functionality. Exercise therapy, including specific methods such as Pilates and trunk stabilization exercises, has been recognized as a safe and effective approach to managing low back pain.

The combination of manual therapy and exercise has been shown to be an effective treatment for low back pain, particularly in chronic cases. Research shows that this multimodal approach significantly improves pain perception, disability and overall functionality in patients suffering from chronic back pain.

In the 2nd group, training in Pain Neuroscience Education (PNE) will be applied. The implementation of the PNE will be done in the form of a short presentation through specific training images. The duration of the PNE will be approximately 5 minutes and will be incorporated into the total time of each session so that each session does not exceed 45 minutes, just like the session time of the 1st intervention group. A total of 6 sessions will be held with the PNE, as many as the total intervention sessions. PNE has emerged as an effective intervention for the management of chronic low back pain.

PNE focuses on teaching patients about how the nervous system works and how pain is created, the difference between acute and chronic pain, the role of the brain in pain perception, and how factors such as stress, hypersensitivity of the nervous system, and beliefs about pain can exacerbate it. The application of PNE can be done before, during or at the end of a physiotherapy intervention. We will apply the PNE before the physiotherapeutic intervention with manual therapy and exercise as it helps in the cognitive preparation of the patient. Educating patients about the mechanisms of pain before physical activity can help reduce movement-related anxiety and fear, promoting a more positive mindset toward rehabilitation. Also, patients who understand their pain have enhanced engagement and are more likely to actively participate in physical interventions, leading to better compliance and outcomes.

Measurements The 60 volunteers of the study, after being approved according to the inclusion criteria, will be randomly divided by lots into 2 groups of 30 people. The 1st group (30 people) will be treated with manual therapy based on Maitland's principles (interview, evaluation, mobilization - mobilization), without any use of physiotherapy machines but with the use of personalized exercises. The 2nd group (30 people) will do the same as group 1 and additional volunteers will participate before, in a Pain Neuroscience Education (PNE) program. The number of sessions that each volunteer will receive will be 6, the duration of each session will be about 45 minutes, the frequency of sessions will be 2 times a week and the total duration of the intervention will be 3 weeks.

Before the start of the interventions (Baseline), the form with the volunteer's demographic and somatometric data will be completed. The volunteer will then be given the self-reported questionnaires mentioned above, in order to complete them on their own. Then the measurement of the range of motion of the lumbar spine with the double inclinometer and the measurement of the pain of the lumbar spine with the mechanical algorithm will be performed.

In between the overall intervention, i.e. before the 4th session, only the questionnaire for the recording of pain will be given.

At the end of the intervention, i.e. after the 6th session, all the self-reported questionnaires given to the baseline will be given again, in order to complete them on their own. The range of motion of the lumbar spine will also be measured again with the double inclinometer and the measurement of the pain of the lumbar spine with the mechanical algometer.

Finally, after 6 months, the volunteers will be contacted by telephone in order to record only their pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be between 18 and 65 years of age,
* the pain in the lumbar region should last for more than 3 months, with at least one attack per week,
* they should not have undergone physiotherapy in the last 6 months prior to the intervention
* have a good knowledge of the Greek language and an adequate level of knowledge, to be informed and sign the consent form and questionnaires

Exclusion Criteria:

* people with clinical conditions that are contraindicated for physiotherapy,
* patients who report red flags,
* people with a history of lumbar surgery,
* people with diagnosed neuromuscular diseases that significantly impair movement,
* people with cardiovascular and respiratory diseases that cause severe shortness of breath or angina
* people with mental disorders, as long as they hinder communication and cooperation with the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | From enrollment to the end of treatment at 3 weeks and after 6 months from the enrollment
  The assessment of pain will be recorded with the Numeric Pain Rating Scale - NPRS questionnaire. "Zero is equivalent to no pain and 10 indicates the worst possible pain."

SECONDARY OUTCOMES:
Disability | From enrollment to the end of treatment at 3 weeks and after 6 months from the enrollment
  The assessment of disability will be recorded with the Oswestry Low Back Pain Disability Index - ODI questionnaire. The ODI questionnaire is a widely recognized patient-reported outcome measure designed to assess the degree of disability in people suffering from low back pain. It consists of 10 questions, which assess various aspects of daily life affected by pain, including personal care, lifting, walking, and social activities.

CONTACTS AND LOCATIONS:
Overall Officials: Zacharias Dimitriadis, Study Director — University of Thessaly

IPD SHARING:
Plan to Share IPD: No